CLINICAL TRIAL: NCT00644033
Title: A Randomized Trial of Frovatriptan for the Intermittent Prevention of Menstrual Migraine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Collaborators: Vernalis (R&D) Ltd (Industry)
Responsible Party: John C. Campbell, Director, Medical Affairs, Endo Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: VML 251 00/02
Record Dates: First submitted 2008-03-24; First posted 2008-03-26 (Estimated); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Menstrually Associated Migraine
MeSH Terms: interventions — frovatriptan

ARMS (3):
- 1 (Active Comparator)
  Interventions: Drug: Frovatriptan
- 2 (Active Comparator)
  Interventions: Drug: Frovatriptan
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Frovatriptan — 2.5 mg tablet administered once daily for 6 days starting 2 days before the anticipated onset of a MAM headache
  Arms: 1
Drug: Frovatriptan — 2.5 mg tablet administered twice daily for 6 days, starting 2 days before the anticipated onset of a MAM headache.
  Arms: 2
Drug: Placebo — placebo tablet administered for 6 days, starting 2 days before the anticipated onset of a MAM headache.
  Arms: 3

SUMMARY:
The primary objective of this study was to determine whether frovatriptan was effective in the prevention of menstrually associated migraine (MAM) headaches when compared to placebo. Secondary objectives included determining the effectiveness of frovatriptan in reducing the incidence, severity and duration of MAM headaches and associated symptoms, to evaluate the safety and tolerability of the two frovatriptan dosing regimens and to compare the effectiveness of these regimens in the prevention of MAM headaches. In this cross-over study, patients treated each of 3 perimenstrual periods (PMPs) with placebo, frovatriptan 2.5 mg daily (QD) and 2.5 mg twice daily (BID) for 6 days, starting 2 days before the anticipated onset of a MAM headache.

A statistically significant reduction in the incidence of MAM headache (p<0.0001) was observed with both dosing regimens of frovatriptan when compared to placebo. Additionally, the frovatriptan BID regimen was superior to the frovatriptan QD regimen in the prevention of MAM headache (p<0.001). Significant reductions in MAM headache severity and duration, the incidence of associated symptoms and characteristics, and the use of rescue medication were observed when the PMP was treated with frovatriptan, compared to placebo. Both dose regimens of frovatriptan were equally well tolerated and no cardiovascular or other safety and tolerability concerns arose with repeated administration of frovatriptan over a 6 day period.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18 years and over
* 12 month or more documented history of menstrual migraine headache, according to International Headache Society classification
* An average frequency of MAM attacks in at lease 3 out of 4 menstrual cycles
* Regular predictable menstrual periods
* Able to accurately predict the onset of MAM headaches occurring between Day -2 and Day +4 of menses
* Able and willing to sign informed consent to comply with study procedures, including completion of diary cards

Exclusion Criteria:

* More than three migraine attacks per month that were not MAM attacks
* Coronary artery disease including coronary vasospasm
* Significant cerebrovascular disease including basilar or hemiplegic migraine
* Uncontrolled hypertension
* Severe hepatic or renal insufficiency
* More than 15 headache days per month
* Any other condition or serious illness which would interfere with optimal participation in the study
* History of clinically relevant allergy, including that to frovatriptan or other triptans
* Pregnant or breast feeding or intending to become pregnant or to breast-feed during study period
* Participated in other frovatriptan menstrual migraine prevention studies
* Use of another investigation drug within 30 days or 5 half-lives (whichever is longer) before the screening visit

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 579 (Actual)
Dates: Start 2001-06; Primary Completion 2002-06 (Actual); Study Completion 2002-06 (Actual)

PRIMARY OUTCOMES:
Incidence of menstrually associated migraine (MAM) headache in the treated peri-menstrual period (PMP)

SECONDARY OUTCOMES:
Incidence of moderate or severe MAM headaches
Incidence of severe MAM headaches
Duration of MAM headaches
Maximum headache intensity
Incidence of MAM headache associated symptoms and characteristics
Duration of MAM headache associated symptoms
Maximum functional impairment score during MAM headache
Incidence of moderate or severe functional impairment during MAM headache
Duration of moderate or severe functional impairment during MAM headache
Incidence of use of rescue medication for the treatment of a MAM headache
Patient satisfaction score at the end of each 6 day treated PMP
Adverse events
Standard hematology and biochemistry
12-lead ECGs, physical exam, vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Elkind, MD, Principal Investigator — Elkind Headache Center
Locations (1):
- Endo Pharmaceuticals, Chadds Ford, Pennsylvania, United States

REFERENCES:
- [Derived] Silberstein SD, Berner T, Tobin J, Xiang Q, Campbell JC. Scheduled short-term prevention with frovatriptan for migraine occurring exclusively in association with menstruation. Headache. 2009 Oct;49(9):1283-97. doi: 10.1111/j.1526-4610.2009.01509.x. Epub 2009 Sep 14. PMID 19751371